CLINICAL TRIAL: NCT00304200
Title: Temodar and Sutent as Therapy for Patients With Malignant Melanoma, a Phase I/II Study
Brief Title: Temodar and Sutent as Therapy for Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding was inadequate to continue; Companies requested closure.
Sponsor: Northern California Melanoma Center (Other)
Collaborators: Pfizer (Industry); Schering-Plough (Industry)
Responsible Party: Lynn E. Spitler, MD, Sponsor/Investigator, Northern California Melanoma Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Temodar/Sutent
Record Dates: First submitted 2006-03-12; First posted 2006-03-17 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Metastatic Malignant Melanoma
Keywords: Metastatic Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm, Open Label (Experimental): Single arm, Open Label Temodar and Sutent
  Interventions: Drug: Temozolomide and SU11248

INTERVENTIONS:
Drug: Temozolomide and SU11248 — First Cohort: Temozolomide 100 mg/m2 orally week 1 and week 3 of a 28-day cycle; SU11248, 25 mg/day orally on weeks 2, 3, and 4 or a 28 day cycle.
  Other Names: Temozolomide is also known as Temodar; SU11248 is also known as Sutent

SUMMARY:
This study is designed to evaluate the safety and appropriate dose of the combination of Temodar and Sutent as first-line therapy for patients with metastatic malignant melanoma (Phase 1). Once the safety and appropriate dose is determined, additional patients will be studied at that dose to determine if there is clinical benefit as determined by the primary end-point of progression-free survival (PFS) at 6 months and additional secondary endpoints (Phase II).

DETAILED DESCRIPTION:
Patients with unresectable metastatic melanoma have a dismal prognosis. The disease responds poorly to currently available chemotherapies and biological agents. The median survival in this patient population is 6 - 10 months and has not improved significantly in decades. The FDA approved DTIC in 1975 and high dose intravenous bolus rIL-2 in 1998 and these are the only agents approved for therapy of patients with metastatic melanoma.

In a Phase III trial reported in 2000, temozolomide (Temodar, Schering-Plough) demonstrated equivalent overall survival to DTIC in patients with metastatic melanoma, and had the advantages of providing improved progression-free survival, ease of administration (oral), and crossing the blood-brain barrier. Temozolomide and DTIC are both precursors of an active metabolite, monomethyl triazenoimidazole carboxamide (MTIC). SU11248 (Sutent, Pfizer) is a multi-targeted receptor tyrosine kinase inhibitor which targets 3 distinct vascular endothelial growth factor receptor (VEGFR-1, -2, and -3), platelet-derived growth factor receptor alpha and beta (PDGFR-α and -β), KIT receptor tyrosine kinases, and fms-related tyrosine kinase 3/Flk2 (FLT3). Although other angiogenic factors have been identified, VEGF is the most potent and specific regulator of angiogenesis and SU11248 targets not just one, but all 3 VEGF signaling pathways. Dacarbazine (DTIC) causes transcriptional up-regulation of VEGF in melanoma cells and this has been postulated as a possible mechanism of escape from chemotherapy efficacy. Temozolomide, which acts through the same metabolite, MTIC, would be expected to have the same activity. PDGFR-α and -β are important new targets in tumor cell proliferation and angiogenesis. PDGF signaling pathways have been implicated in the development and growth of solid tumors. Inhibition of PDGF receptors has been shown to inhibit angiogenesis, tumor vascular maturation and maintenance, and tumor cell proliferation - inducing tumor regression. In a murine model, the combination of chemotherapy with VEGF and PDFG receptor inhibitors resulted in a remarkable survival advantage.

The study is an open-label, single arm trial. The patient sample will be approximately 56-62 individuals, males and females 18 years of age or older with measurable metastatic melanoma. Study participants must meet a number of laboratory criteria in order to be admitted into the study. The study duration is expected to be approximately 2 years. Patients will be offered treatment for up to 1 year and are expected to complete a median of 6 cycles of treatment.

An interim analysis of safety will be conducted after completion of treatment of 6 patients in each cohort and a determination will be made as to whether or not to continue to the next cohort according to the specifications in the protocol. If an acceptable dosing regimen is found, the study will proceed to a Phase II portion. Progression-free survival will be determined for the 6 month time point when all patients have completed the study. The study has ≥90% power to detect an increase in the 6-month progression-free survival rate from ≤15%, the result expected for patients receiving available first-line therapy, to ≥35% for patients receiving the combination of temozolomide and SU11248, based on a one group chi-square test with a 0.05 two-sided significance level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed, (surgically incurable or unresectable)stage IV metastatic malignant melanoma.
* Patients must not have received any prior cytokine or chemotherapy for stage IV disease.
* ECOG performance status of 0-1.
* Age greater than or equal to 18 years.
* Adequate hematologic, renal and liver function as defined by laboratory values performed within 28 days prior to initiation of dosing.

  * Absolute neutrophil count (ANC) greater than or equal to 1500/uL
  * Platelet count greater than or equal to 100,000/uL
  * Hemoglobin greater than or equal to 10.0 g/dL
  * Serum creatinine ≤ 1.5 upper limit of laboratory normal
  * Total serum bilirubin less than or equal to1.5 times upper limit of laboratory normal
  * LDH less than or equal to 2 times upper limit of laboratory normal
  * Serum aspartate transaminase (ASAT/SGOT) or serum alanine transaminase (ALAT/SGPT) ≤ 2.5 times upper limit of laboratory normal, and ≤ 5 times upper limit of laboratory normal in cases of liver metastasis
* Patients must have recovered from effects of major surgery.
* Women of childbearing potential should be using an effective method of contraception. Women of childbearing potential must have a negative urine or serum pregnancy test up to 28 days prior to commencement of dosing and be practicing medically approved contraceptive precautions for at least 6 months after completion of treatment as directed by their physician.
* Men should use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before trial entry.
* Before study entry, written informed consent must be obtained. Written informed consent must be obtained from the patient prior to performing any study-related procedures.

Exclusion Criteria:

* Major surgery or radiation therapy within 4 weeks of starting the study treatment.
* Evidence of brain metastases.
* NCI CTCAE Version 3.0 grade 3 hemorrhage within 4 weeks of starting the study treatment.
* History of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade equal to or greater than 2.
* Prolonged QTc interval on baseline EKG.
* Uncontrolled hypertension (>150/100 mm Hg despite optimal medical therapy).
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Known active infection.
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Treatment with drugs with dysrhythmic potential including terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, and/or indapamide.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Frequent vomiting or medical condition which could interfere with oral medication intake (e.g. partial bowel obstruction).
* Previous cancer (unless a DRS interval of at least 5 years) or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin.
* Known clinically uncontrolled infectious disease including HIV positivity or AIDS-related illness.
* Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of this combination | March 2006 through October 2007
Determine the Maximum Tolerated Dose (MTD) of this combination | March 2006 through October 2007

SECONDARY OUTCOMES:
Progression-free survival (PFS) at 6 months | March 2006 through October 2007
Progression-free survival (PFS) | March 2006 through October 2007
Overall survival (OS) | October 2006 through January 2009
Objective Response Rate (RR)in patients with measurable lesions | March 2006 through October 2007
Duration of Objective Response in patients with measurable lesions | March 2006 through October 2007
Correlation of outcome with MGMT promoter methylation | March 2006 through October 2007

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E. Spitler, MD, Principal Investigator — Northern California Melanoma Center
Locations (1):
- Northern California Melanoma Center, San Francisco, California, United States

REFERENCES:
- [Background] Middleton MR, Grob JJ, Aaronson N, Fierlbeck G, Tilgen W, Seiter S, Gore M, Aamdal S, Cebon J, Coates A, Dreno B, Henz M, Schadendorf D, Kapp A, Weiss J, Fraass U, Statkevich P, Muller M, Thatcher N. Randomized phase III study of temozolomide versus dacarbazine in the treatment of patients with advanced metastatic malignant melanoma. J Clin Oncol. 2000 Jan;18(1):158-66. doi: 10.1200/JCO.2000.18.1.158. PMID 10623706
- [Background] Hicklin DJ, Ellis LM. Role of the vascular endothelial growth factor pathway in tumor growth and angiogenesis. J Clin Oncol. 2005 Feb 10;23(5):1011-27. doi: 10.1200/JCO.2005.06.081. Epub 2004 Dec 7. PMID 15585754
- [Background] Lev DC, Ruiz M, Mills L, McGary EC, Price JE, Bar-Eli M. Dacarbazine causes transcriptional up-regulation of interleukin 8 and vascular endothelial growth factor in melanoma cells: a possible escape mechanism from chemotherapy. Mol Cancer Ther. 2003 Aug;2(8):753-63. PMID 12939465
- [Background] George D. Targeting PDGF receptors in cancer--rationales and proof of concept clinical trials. Adv Exp Med Biol. 2003;532:141-51. doi: 10.1007/978-1-4615-0081-0_12. PMID 12908555
- [Background] Bergers G, Song S, Meyer-Morse N, Bergsland E, Hanahan D. Benefits of targeting both pericytes and endothelial cells in the tumor vasculature with kinase inhibitors. J Clin Invest. 2003 May;111(9):1287-95. doi: 10.1172/JCI17929. PMID 12727920
- [Background] Erber R, Thurnher A, Katsen AD, Groth G, Kerger H, Hammes HP, Menger MD, Ullrich A, Vajkoczy P. Combined inhibition of VEGF and PDGF signaling enforces tumor vessel regression by interfering with pericyte-mediated endothelial cell survival mechanisms. FASEB J. 2004 Feb;18(2):338-40. doi: 10.1096/fj.03-0271fje. Epub 2003 Dec 4. PMID 14657001
- [Background] Pietras K, Hanahan D. A multitargeted, metronomic, and maximum-tolerated dose "chemo-switch" regimen is antiangiogenic, producing objective responses and survival benefit in a mouse model of cancer. J Clin Oncol. 2005 Feb 10;23(5):939-52. doi: 10.1200/JCO.2005.07.093. Epub 2004 Nov 22. PMID 15557593